CLINICAL TRIAL: NCT04332640
Title: Clinical Investigation of the Next Generation Phaco System (VERITAS Vision System)
Brief Title: Clinical Evaluation of the Next Generation Phaco System
Acronym: ALPINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALPI-101-SYST
Record Dates: First submitted 2020-04-01; First posted 2020-04-02 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Next Generation Phaco System (Experimental): VERITAS Vision System
  Interventions: Device: VERITAS Vision System

INTERVENTIONS:
Device: VERITAS Vision System — The investigators or designees will perform routine small-incision cataract surgery via phacoemulsification and use the VERITAS Vision system. The Investigator or designee will then complete a questionnaire regarding the clinical use of the VERITAS Vision system. The system log files automatically generated by the VERITAS Vision system after completion of each surgery will be collected.

SUMMARY:
This study is a prospective, open-label clinical study of the VERITAS Vision System.

The study will be conducted at up to three sites, with minimum 55 eyes and up to 150 eyes to be treated. The investigator or designee will perform the cataract surgery with the VERITAS Vision System on the subjects. The data from the system log files, the questionnaire, the operative report and other medical records will be used to assess the clinical utilization of the VERITAS Vision System.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age.
* Cataracts for which cataract extraction and posterior chamber IOL implantation have been planned.
* Availability, willingness, ability and sufficient cognitive awareness to comply with study requirements, examination procedures, and visits.
* Be willing to provide informed consent and authorization to disclose protected health information or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical procedures in the governing countries.

Exclusion Criteria:

* Expected surgical difficulties at the time of cataract extraction, which may increase the potential for complications (e.g., persistent bleeding, significant iris damage, uncontrolled intraocular pressure change, or significant vitreous prolapse or loss).
* Subjects with only one good eye (e.g. amblyopic condition etc.).
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration, including pseudoexfoliation, trauma, or posterior capsule defects.
* History or current use of alpha-1 antagonist medication (e.g., Flomax).
* Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study or for which cataract surgery is contraindicated.
* Pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils).
* Is pregnant, or is breast feeding, or intend to become pregnant during the study.
* Concurrent participation or expected participation in an interventional (i.e., surgical or pharmaceutical interventional) clinical trial within 14 days prior to study screening.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trial, Study Director — Johnson & Johnson Surgical Vision
Locations (2):
- ACE Eyecare, Inc, Bakersfield, California, United States
- Grupo Oftalmo & Plastico, Centro de Oftalmologia y Cirugia Plastica, El Escalón, San Salvador Department, El Salvador

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 115 eyes of 79 subjects were enrolled and treated at 2 sites by 6 investigators. Of these 79 subjects (115 eyes) , 36 subjects had bilateral (72 eyes) surgeries and 43 subjects had unilateral (43 eyes) surgeries.
Units Other Than Participants: Eyes
Groups:
- Veritas Vision System: Next Generation Phaco System
Period: Overall Study
Arm/Group | Veritas Vision System
Started | 79; 115 Eyes
Completed | 79; 115 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | Veritas Vision System
Number analyzed (Participants) | 79
Age, Customized [Number; unit: Participants]
  <30 years | 0
  30-39 years | 0
  40-49 years | 2
  50-59 years | 17
  60-69 years | 32
  >=70 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2
  Black | 0
  Native Hawaiian/Pacific Islander | 0
  Caucasian | 36
  Central and South American | 41
  Other race | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Surgeon Satisfaction Rating Score of 4 or 5
Description: Surgeons rated the following Questionnaire items regarding satisfaction with the VERITAS Vision System, using 1 - 5 scale (acceptability considered favorable for scores of 4 and 5, where 4 is Satisfied and 5 is Very Satisfied)
Time Frame: 1 day postoperative
Population: All Eyes treated with Veritas Vision System
  * 1 Surgeon rating was disqualified in Overall satisfaction with VERITAS Vision System, making N=114
Measure: Number (95% Confidence Interval); unit: Proportion of Eyes
Units Other Than Participants: Eyes
Groups:
- Veritas Vision System: n/N (Eyes with ratings of 4 or 5/eyes treated)
Arm/Group | Veritas Vision System
Number analyzed (Participants) | 79
Number analyzed (Eyes) | 115
Proportion of Eyes
  Rating of overall satisfaction with anterior chamber stability | 0.991 [.95 to 1.00]
  Rating of followability | 0.991 [0.95 to 1.00]
  Rating of holdability | 0.991 [0.95 to 1.00]
  Rating of Phaco (cutting) efficiency | 1.00 [0.97 to 1.00]
  Satisfaction with usability of VERITAS Vision System | 1.00 [0.97 to 1.00]
  Overall satisfaction with VERITAS Vision System *: number analyzed (Eyes) | 114
  Overall satisfaction with VERITAS Vision System * | 0.991 [0.95 to 1.00]

ADVERSE EVENTS:
Time Frame: 48 days
Description: Analysis population include all 79 participants treated using the VERITAS Vision System. All adverse events (AEs), ocular and non-ocular, were monitored/assessed and planned to be reported for each eye separately.
Arm/Group | Veritas Vision System
All-Cause Mortality (participants affected / at risk) | 0/79
Serious Adverse Events (participants affected / at risk) | 1/79
Other Adverse Events (participants affected / at risk) | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veritas Vision System (N=79)
Posterior capsule rupture due to surgeon error (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime.

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT04332640/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT04332640/SAP_001.pdf